CLINICAL TRIAL: NCT03349645
Title: An Open Label Extension Study to Assess the Safety of Long-Term Treatment With a 4 mL Intra-Articular Injection of Ampion in Adults With Pain Due to Severe Osteoarthritis of the Knee
Brief Title: Open Label Extension to Assess the Safety of Long-Term Treatment With Ampion for Severe Osteoarthritis (OA) of the Knee
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated by Sponsor due to absence of significant safety findings.
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AP-003-C-OLE
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Results first posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-08

CONDITIONS: Severe Osteoarthritis of the Knee
Keywords: Osteoarthritis; osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMPION™ 4 mL dose (Experimental): 4 mL intra-articular injection of AMPION™
  Interventions: Biological: 4 mL injection of AMPION™

INTERVENTIONS:
Biological: 4 mL injection of AMPION™ — 4 mL injection of AMPION™

SUMMARY:
This Open Label Extension (OLE) study will assess the safety of long-term treatment with a 4 mL intra-articular injection of Ampion™ in adults with pain due to severe osteoarthritis of the knee

DETAILED DESCRIPTION:
An Open Label Extension (OLE) study will assess the safety of long-term treatment with a 4 mL intra-articular injection of Ampion™ in adults with pain due to severe osteoarthritis of the knee.

The primary trial objective was to evaluate the safety of a 4-mL intra-articular (IA) injection of Ampion with repeat dosing every 12 weeks for 52 weeks with five total injections of Ampion.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who completed the AP-003-C Main study and have not developed any exclusionary criteria
2. Able to provide written informed consent to participate in the study
3. Willing and able to comply with all study requirements and instructions of the site study staff
4. Male or female, 40 years to 85 years old (inclusive), as assessed in the AP-003-C Main Study
5. Must be ambulatory, as assessed in the AP-003-C Main Study
6. Study knee must have a clinical diagnosis of OA and supported by radiological evidence (Kellgren Lawrence Grade IV) as assessed in the AP-003-C Main Study.
7. Moderate to moderately-severe OA pain in the study knee (rating of at least 1.5 on the WOMAC Index 3.1 5-point Likert Pain Subscale), as assessed in the AP-003-C Main Study
8. Moderate to moderately-severe OA function in the study knee (rating of at least 1.5 on the WOMAC Index 3.1 5-point Likert Function Subscale), as assessed in the AP-003-C Main Study
9. WOMAC A, 5-point Likert pain subscale <1.5 in the contralateral knee, as assessed in the AP-003-C Main Study
10. Ability to discontinue NSAID ± 72 hours before/after injections (in-office visits). Low-dose Aspirin (81 mg) is allowed during the study but must not be taken at least 24 hours prior to in-office visits.
11. No analgesia (including acetaminophen [paracetamol]) taken 24 hours prior to an efficacy measure

Exclusion Criteria:

1. As a result of medical review and screening investigation, the Principal Investigator considers the patient unfit for the study
2. Known clinically significant liver abnormality (e.g., cirrhosis, transplant, etc.)
3. A history of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin is not an exclusion criterion)
4. A history of allergic reactions to excipients in 5% human albumin (N-acetyltryptophan, sodium caprylate)
5. Presence of tense effusions
6. Inflammatory or crystal arthropathies, acute fractures, history of aseptic necrosis or joint replacement in the affected knee
7. Isolated patella femoral syndrome, also known as chondromalacia
8. Any other disease or condition interfering with the free use and evaluation of the index knee for the duration of the trial (e.g. cancer, congenital defects, spine osteoarthritis)
9. Major injury to the index knee within the last 12 months
10. Severe hip osteoarthritis ipsilateral to the index knee
11. Any pain that could interfere with the assessment of study knee pain (e.g. pain in any other part of the lower extremities, pain radiating to the knee)
12. Any pharmacological or non-pharmacological treatment targeting OA started or changed 4 weeks prior to entry into the OLE study, or likely to be changed during the duration of the OLE study
13. Pregnancy or planning to become pregnant during the study
14. Use of the following medications:

    1. No IA injected pain medications in the study knee during the study. No Hyaluronic Acid (HA) or steroid injections in the study knee at least 12 weeks prior to Day 84 of the Extension Study. HA and steroid injections in the contralateral knee (non-study knee) are acceptable while on study except ± 14 days of an Ampion injection in the study knee.
    2. No analgesics containing opioids
    3. NSAIDs are not permitted ± 72 hours before/after injections at in-office visits; acetaminophen is available as a rescue medication during the study from the provided supply
    4. No topical treatment on the study knee during the study
    5. No significant anticoagulant therapy (e.g. Heparin or Lovenox) during the study (treatment such as Aspirin and Plavix are allowed)
    6. No systemic treatments that may interfere with safety or efficacy assessments during the study
    7. No immunosuppressants
    8. No use of corticosteroids
    9. No human albumin treatment in the 3 months prior to the AP-003-C Main Study or interim period prior to enrollment into the OLE study. No human albumin treatment throughout the duration of the OLE study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, MD, Study Director — Ampio Pharmaceuticals. Inc.
Locations (11):
- United States (11):
  - Central Research Associates, Inc., Birmingham, Alabama
  - CORE Orthopaedic Medical Center, Encinitas, California
  - St. Joseph Heritage, Fullerton, California
  - Westlake Medical Research, Thousand Oaks, California
  - Drug Studies America, Marietta, Georgia
  - Healthcare Research Netword, Blue Island, Illinois
  - Heartland Research Associates, Wichita, Kansas
  - Healthcare Network Research, Hazelwood, Missouri
  - Coastal Carolina Center at Lowcountry Orthopaedics, North Charleston, South Carolina
  - Tekton Research, Austin, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who had completed clinical trial AP-003C were eligible to enroll in the open label extension study. All subjects were assigned to the Ampion treatment group.
Pre-assignment Details: No pharmacological or non-pharmacological treatment targeting osteoarthritis (OA) started or changed 4 weeks prior to entry into the study, or likely to be changed during the duration of the study
Groups:
- Ampion 4 mL Dose: 4 mL Ampion (<5 kilodalton (kDa) ultrafiltrate of 5% Human Serum Albumin (HSA)), solution
Period: Overall Study
Arm/Group | Ampion 4 mL Dose
Started | 94
Completed | 12
Not Completed | 82
Not completed — Sponsor Terminated Study | 75
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 1
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ampion 4 mL Dose
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 89
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 66
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 94

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs)
Description: Incidence and severity of treatment emergent adverse events (TEAEs) evaluated up to 52 weeks, including the 12 weeks in the Main study AP-003-C (NCT03182686).
Time Frame: 52 weeks
Population: Intent To Treat (ITT)
Measure: Number; unit: Events
Arm/Group | Ampion 4 mL Dose
Number analyzed (Participants) | 94
Events
  Mild treatment-emergent adverse event (TEAE) | 21
  Moderate treatment-emergent adverse event (TEAE) | 11
  Severe treatment-emergent adverse event (TEAE) | 2

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: Patients will be followed for the occurrence of AEs up to 52 weeks, including the 12 weeks in the Main study AP-003-C (NCT03182686).
Arm/Group | Ampion 4 mL Dose
All-Cause Mortality (participants affected / at risk) | 0/94
Serious Adverse Events (participants affected / at risk) | 0/94
Other Adverse Events (participants affected / at risk) | 22/94
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ampion 4 mL Dose (N=94)
Non-Alcoholic Fatty Liver (Hepatobiliary disorders) | 2
Tooth Fracture (Injury, poisoning and procedural complications) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Joint Crepitation (Musculoskeletal and connective tissue disorders) | 2
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT03349645/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/45/NCT03349645/SAP_001.pdf